CLINICAL TRIAL: NCT02995694
Title: Clinical Endpoint Therapeutic Equivalence Multi-Site Study Comparing Estradiol Vaginal Cream (0.01%; Alvogen Pine Brook LLC.) to Estrace® Cream (0.01%; Warner Chilcott) in Postmenopausal Females With Atrophic Vaginitis
Brief Title: A Study Comparing Estradiol Vaginal Cream to Estrace® Cream in Females With Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvogen Pine Brook LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 71462901
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test (Experimental): Estradiol Vaginal Cream
  Interventions: Drug: Estradiol
- Reference. (Active Comparator): Estrace Vaginal Cream
  Interventions: Drug: Reference
- Placebos (Placebo Comparator): Placebo with no active pharmaceutical ingredients. Topical vaginal cream
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Estradiol — Estradiol Vaginal Cream
  Other Names: Estadiol Vaginal Cream
  Arms: Test
Drug: Placebos — Placebo with no active pharmaceutical ingredients. Topical vaginal cream
  Other Names: Topical Vaginal Cream
  Arms: Placebos
Drug: Reference — Estrace Vaginal Cream
  Other Names: Topical Vaginal Cream
  Arms: Reference.

SUMMARY:
The purpose of this study is to determine the therapeutic equivalence of Alvogen's estradiol vaginal cream to Estrace® cream and superiority of both products to placebo. The protocol describes a randomized, double-blind, multi-dose, placebo-controlled, parallel study of a 7 day treatment.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, parallel group, multiple-site study was designed to evaluate the therapeutic efficacy and safety of a generic Estradiol Vaginal Cream USP, 0.01% (Alvogen Pine Brook LLC) compared to the FDA Reference Listed Drug (RLD), Estrace® (estradiol vaginal cream USP, 0.01%, Warner Chilcott) in patients with atrophic vaginitis. Additionally, both the Test and the RLD formulations were tested for superiority against a Placebo.

Following the 14-day screening period, patients who continued to meet the inclusion/exclusion criteria were randomized in a 2:2:1 ratio (Test: Reference: Placebo) for 7 days of treatment.

Five hundred and thirty-five (535) patients were randomized to one of the three study products as follows:

* Test: Estradiol Vaginal Cream USP, 0.01% (Alvogen Pine Brook LLC)
* Reference: Estrace® (estradiol vaginal cream USP, 0.01%) (Warner Chilcott)
* Placebo: Test product vehicle cream (Alvogen Pine Brook LLC)

Patients completed up to three clinic visits as follows:

* Visit 1 - Screening: Day -14 to Day -1
* Visit 2 - Randomization: Day 1
* Visit 3 - End of Study: Day 8, maximum Day 10

Study product was self-administered by the patient for 7 days according to the dosing instructions provided. Each patient was required to dose once daily at approximately the me of day for 7 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent that meets all criteria of current FDA regulations
2. Females age: 30-75 years old inclusive who are postmenopausal.
3. Postmenopausal defined as at least 12 months of spontaneous amenorrhea or at least 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or at least 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy. Hysterectomy without oophorectomy if of age that investigator believes would have naturally reached 12 months of spontaneous amenorrhea.
4. Baseline evaluation requirements:

   * ≤5% superficial cells on vaginal smear cytology
   * Vaginal pH > 5.0
   * At least one patient self-assessed moderate to severe symptom of vulvar and/or vaginal atrophy (VVA) from the following list that is identified by the subject:
   * Vaginal dryness
   * Vaginal and/or vulvar irritation/itching
   * Dysuria
   * Vaginal pain associated with sexual activity*
   * Vaginal bleeding associated with sexual activity (absence vs. presence)* *provided that patient is currently sexually active and plans to remain so throughout study.
5. Normal breast exam at screening and mammogram completed within 9 months prior to screening in patients >40 years old.
6. For women with an intact uterus, an endometrial thickness < 4 mm as determined by vaginal ultrasonography.
7. Documented PAP smear conducted within previous 12 months with no findings that the Investigator believes would contraindicate the use of topical vaginal estradiol

Exclusion Criteria:

1. Females younger than 30 years of age or older than 75 years of age
2. Patients with a serum FSH level of ≤ 40mIU/ml at screening.
3. Greater than 5% superficial cells on vaginal cytology.
4. Vaginal pH ≤ 5
5. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder (including significant liver/kidney impairment) or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
6. Patients with an intact uterus should have vaginal ultrasonography results to confirm an inactive endometrial lining. Patients with an endometrial thickness equal to or greater than 4mm should be excluded.
7. Patients with known, suspected or current history of carcinoma of the breast. All patients over the age of 40 must have had a mammogram performed within 9 months of the study start and all patients will have a physical breast exam performed at screening.
8. Patients with baseline systolic blood pressure of > 150mm Hg and/or diastolic pressure > 90 mm Hg
9. Any patient with undiagnosed vaginal bleeding or significant risk factors for endometrial cancer.
10. Any history of estrogen-dependent neoplasia (e.g., endometrial cancer).

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meena Venugopal, Ph.D., Study Chair — Alvogen Pine Brook LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test | Reference. | Placebos
Started | 215 | 211 | 109
Completed | 181 | 183 | 94
Not Completed | 34 | 28 | 15

BASELINE CHARACTERISTICS:
Groups:
- Estradiol Vaginal Cream: Estradiol Vaginal Cream, 0.01%, administered once daily for 7 days. Estradiol Vaginal Cream, 0.01%: Estradiol Vaginal Cream, 0.01% (1 x 2 g for 7 days)
- Estrace Vaginal Cream: Estrace Vaginal Cream, 0.01%, administered once daily for 7 days. Estrace Vaginal Cream, 0.01%: Estradiol Vaginal Cream, 0.01% (1 x 2 g for 7 days)
- Placebo: Placebo Cream, administered once daily for 7 days. Placebo Cream, (1 x 2 g for 7 days)
- Total: Total of all reporting groups
Arm/Group | Estradiol Vaginal Cream | Estrace Vaginal Cream | Placebo | Total
Number analyzed (Participants) | 181 | 183 | 94 | 458
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 167 | 172 | 89 | 428
  >=65 years | 14 | 11 | 5 | 30
Age, Continuous [Mean (Full Range); unit: years] | 59.0 [42 to 75] | 59.4 [45 to 74] | 59.9 [47 to 74] | 59.4 [42 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 183 | 94 | 458
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 67 | 30 | 159
  Not Hispanic or Latino | 119 | 116 | 64 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 25 | 7 | 46
  White | 165 | 155 | 85 | 405
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 181 | 183 | 94 | 458

OUTCOME MEASURES:

1. Primary Outcome: Vaginal Cytology
Description: Number of patients in PP population identified as responders at end of the study.
Time Frame: Day 8
Measure: Number; unit: participants
Arm/Group | Test | Reference. | Placebos
Number analyzed (Participants) | 181 | 183 | 94
participants | 29 | 19 | 0

2. Secondary Outcome: Patient Self-assessment of the Symptoms of Vulvar and Vaginal Atrophy
Description: Number of participants with the most bothersome vulvar and/or vaginal atrophy symptom treatment success at end of study. A "Treatment Success" was defined as a score of 0 or 1 at Day 8 (maximum Day 10) for the symptom identified at baseline as the most bothersome. This evaluation was based on patient self-assessed symptoms of VVA on a scale of 0 to 3 where 0 = none, 1 = mild, 2 = moderate, and 3 = severe.
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo arm
Arm/Group | Estradiol Vaginal Cream | Reference | Placebo
Number analyzed (Participants) | 181 | 183 | 94
Participants | 115 | 114 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Description: There was one SAE, a death, reported for a subject during screening who had not yet been randomized into the study.
Arm/Group | Test | Reference. | Placebos
All-Cause Mortality (participants affected / at risk) | 0/215 | 0/211 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/215 | 0/211 | 0/109
Other Adverse Events (participants affected / at risk) | 88/215 | 85/211 | 30/109
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=215) | Reference. (N=211) | Placebos (N=109)
Gastrointestinal (Gastrointestinal disorders) | 36 | 36 | 20
Breast Tenderness (Reproductive system and breast disorders) | 36 | 37 | 5
Nervous System Disorders (Nervous system disorders) | 13 | 19 | 5
Psychiatric disorders (Psychiatric disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days